CLINICAL TRIAL: NCT04446208
Title: Endoscopic Treatment of Post-operative Fistula of the Upper Digestive Tract
Brief Title: Endoscopy for Post-operative Fistula
Acronym: FISTULENDO
Status: Completed | Type: Observational
Sponsor: Aymeric Becq (Other)
Responsible Party: Sponsor-Investigator, Aymeric Becq, Medical doctor-principal Investigator, French Society of Digestive Endoscopy
Organization: French Society of Digestive Endoscopy (Other)
Other Study IDs: SFED N 146
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Post-operative Fistula
Keywords: Fistula; Upper digestive tract; Cancer
MeSH Terms: conditions — Fistula; Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopy — Endoscopic treatment will consist in placement of a metal stent in a patient with early fistula (< 15 days) and/or a large fistula orifice, and no abscess, or double pigtail plastic stents if the fistula is older than 15 days and the orifice is small.

SUMMARY:
Endoscopic treatment of early post-operative fistula in patients with underlying esophageal or gastric cancer has now become the standard of care. However, data regarding the yield of this type of treatment is lacking. This study aims to evaluate endoscopic management of this post-operative complication. The main outcome of this prospective observational study conducted in tertiary centers in France is fistula healing defined as the absence of collection on CT scan (with opacification) in a patient on PO diet, 3 months after the end of the endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Early fistula (< 30 days)
* Post surgery: Lewis Santy, Akiyama, partial or total gastrectomy
* Indication of endoscopic management: metal stents and/or plastic stents

Exclusion Criteria:

* Pregnancy
* Incapable of decision making and informed consent
* Life expectancy < 1 month
* General anesthesia contra-indication
* Late fistula (> 30 days)
* Prior endoscopic treatment
* Wall ischemia
* Duodenum or small bowel fistula
* Post bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with post-operative fistula of the upper digestive tract, in the setting of a cancerous underlying condition.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
fistula healing | 3 months after the end of the endoscopic
  The main outcome is fistula healing defined as the absence of collection on CT scan (with opacification) in a patient on PO diet, 3 months after the end of the endoscopic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Antoine Hospital, Paris, France